CLINICAL TRIAL: NCT03528642
Title: A Phase 1b Trial of Telaglenastat (CB-839) HCI in Combination With Radiation Therapy and Temozolomide in Patients With IDH-Mutated Diffuse Astrocytoma and Anaplastic Astrocytoma
Brief Title: Telaglenastat With Radiation Therapy and Temozolomide in Treating Patients With IDH-Mutated Diffuse Astrocytoma or Anaplastic Astrocytoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-00876; NCI-2018-00876 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10218 (Other: Dana-Farber - Harvard Cancer Center LAO); 10218 (Other: CTEP); UM1CA186686 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2018-05-17; First posted 2018-05-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Astrocytoma, IDH-Mutant, Grade 2; Astrocytoma, IDH-Mutant, Grade 3
MeSH Terms: conditions — Astrocytoma; Lymphoma, Follicular | interventions — Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (telaglenastat, temozolomide, RT) (Experimental): Patients receive telaglenastat PO BID 7 days a week, temozolomide PO QD 7 days a week, and undergo RT 5 days a week for up to 5.5 weeks (diffuse astrocytoma) or 6.5 weeks (anaplastic astrocytoma) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Telaglenastat Hydrochloride; Drug: Temozolomide

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Telaglenastat Hydrochloride — Given PO
  Other Names: CB-839 HCl; Glutaminase Inhibitor CB-839 Hydrochloride
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase 1b trial studies the side effects and best dose of telaglenastat in combination with radiation therapy and temozolomide in treating patients with IDH-mutated diffuse or anaplastic astrocytoma. Telaglenastat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving telaglenastat with radiation therapy and temozolomide may work better than surgery, radiation therapy, and temozolomide in treating patients with IDH-mutated diffuse astrocytoma or anaplastic astrocytoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D) of telaglenastat (CB-839) hydrochloride (HCl) when combined with radiation therapy (RT) and temozolomide (TMZ) in patients with newly diagnosed IDH-mutated diffuse astrocytoma (DA) and anaplastic astrocytoma (AA).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. Determine the safety and tolerability of RT/TMZ/telaglenastat (CB-839) HCl in patients based on physician reported adverse event (AE) data.

III. Estimate the 2-year progression-free survival (PFS2) of RT/TMZ/telaglenastat (CB-839) HCl in patients with IDH-mutated glioma based on the Response Assessment in Neuro-Oncology (RANO) criteria.

IV. Estimate the 2-year overall survival (OS2) of RT/TMZ/telaglenastat (CB-839) HCl in patients with IDH-mutated glioma based on RANO criteria.

CORRELATIVE OBJECTIVES:

I. Determine the minor response rate (MRR) and clinical benefit rate (CBR) for the combination of telaglenastat (CB-839) HCl and RT/TMZ in IDH-mutated glioma based on RANO criteria.

II. Determine the patient-reported tolerability of RT/TMZ/telaglenastat (CB-839) HCl using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) instrument to measure self-reported symptom severity and interference with daily activities.

II. Determine the neurocognitive impact of telaglenastat (CB-839) HCl when used in combination with RT/TMZ.

III. Determine the effect of telaglenastat (CB-839) HCl/RT/TMZ on plasma oncometabolite levels of glutamine, glutamate, aspartate, asparagine, and 2-hydroxyglutarate (2-HG) in patients with IDH-mutated glioma and associate the changes with disease response.

IV. Determine the effect of telaglenastat (CB-839) HCl/RT/TMZ on tumor glutamine and glutamate MRS signals in patients with IDH-mutated glioma and associate the signal with disease response.

V. Determine the pharmacokinetics (PK) of telaglenastat (CB-839) HCl when used alone and in combination with TMZ.

VI. To perform molecular profiling assays on archived tumor tissue and peripheral blood, including, but not limited to, low-pass whole genome sequencing (WGS), whole exome sequencing (WES), and messenger ribonucleic acid (RNA) sequencing (RNA-Seq) in order to VIa. Identify potential predictive and prognostic biomarkers beyond any genomic alteration by which treatment may be assigned.

VIb. Identify resistance mechanisms using genomic deoxyribonucleic acid (DNA)- and RNA-based assessment platforms.

VII. To contribute genetic analysis data from de-identified biospecimens to Genomic Data Commons (GDC), a well annotated cancer molecular and clinical data repository, for current and future research; specimens will be annotated with key clinical data, including presentation, diagnosis, staging, summary treatment, and if possible, outcome.

VIII. To bank formalin-fixed, paraffin-embedded (FFPE) tissue, blood (for cell-free DNA analysis), and nucleic acids obtained from patients at the Experimental Therapeutics Clinical Trials Network (ETCTN) Biorepository at Nationwide Children's Hospital.

OUTLINE: This is a dose escalation study of telaglenastat.

Patients receive telaglenastat orally (PO) twice daily (BID) 7 days a week, temozolomide PO once daily (QD) 7 days a week, and undergo RT 5 days a week for up to 5.5 weeks (diffuse astrocytoma) or 6.5 weeks (anaplastic astrocytoma) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologic or molecular confirmation of either IDH-mutant DA or IDH-mutant AA. Acceptable IDH mutations for study eligibility include any IDH1 mutation at codon 132 or any IDH2 mutation at codon 172.
* Age >= 16 years. The intended neurocognitive tests have not been validated in children below the age of 16.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%).
* Hemoglobin > 9.0 g/dL (within 14 days prior to registration)
* Leukocytes >= 3.0 x 10^9/L (within 14 days prior to registration)
* Absolute neutrophil count >= 1.5 x 10^9/L (within 14 days prior to registration)
* Platelets >= 100 x 10^9/L (within 14 days prior to registration)
* International normalized ratio (INR) =< 1.5 x upper limit of normal (ULN) (within 14 days prior to registration)
* Partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) =< 1.5 x ULN (within 14 days prior to registration)
* Patients on a stable dose of anti-coagulation therapy will be allowed to participate if they have no signs of bleeding or clotting and the INR/PT and PTT/aPTT results are compatible with an acceptable risk-benefit ratio as per the investigator's discretion.
* Total bilirubin =< 1.5 x institutional ULN and < 3 mg/dL for patients with Gilbert's disease (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) & alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (within 14 days prior to registration)
* Creatinine =< 1.5 x institutional ULN or creatinine clearance >= 60 mL/minute
* If there is history of human immunodeficiency virus (HIV) infection, patients must be on effective antiretroviral therapy and HIV viral load must be undetectable within 6 months of study enrollment.
* If there is history of chronic hepatitis B virus (HBV) infection, patients must have either been treated or are on suppressive therapy (as indicated), and HBV viral load must be undetectable.
* If there is history of hepatitis C virus (HCV) infection, patients must have been treated and HCV viral load must be undetectable.
* Patient must have measurable disease by RANO criteria (dose expansion cohort only).
* Patient must be at least 7 days beyond stereotactic biopsy and/or at least 14 days beyond open craniotomy at the time of registration.
* Patients must have been on a stable or decreasing dose of corticosteroids over the last 7 days at the time of registration.
* Patients must have been on a stable or decreasing dose of antiepileptic therapy over the last 14 days at the time of registration.
* Females of childbearing potential must have a negative pregnancy test (=< 14 days) prior to start of trial treatment. The effects of telaglenastat (CB-839) HCl on the developing human fetus are unknown. For this reason and because alkylating agents as well as TMZ are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of telaglenastat (CB-839) HCl administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better.
* Availability of archival FFPE tumor tissue collected within 12 months prior to registration.

Exclusion Criteria:

* Patients must not have received prior chemotherapy to treat the glioma.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to telaglenastat (CB-839) HCl or TMZ.
* Patient must not have received prior radiation therapy to the brain. Prior radiation therapy to the head and neck is also excluded if radiation fields overlap.
* No prior use of Gliadel wafers.
* Patient must have no evidence of either infratentorial or spinal involvement with tumor.
* Patients who are unable to swallow tablets.
* Patients who are at risk for impaired absorption of oral medication including, but not limited to, refractory vomiting, gastric resection/bypass, and duodenal/jejunal resection.
* Patients with uncontrolled intercurrent illness.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for more than 3 years.
* Pregnant women are excluded from this study because telaglenastat (CB-839) HCl is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with telaglenastat (CB-839) HCl, breastfeeding should be discontinued if the mother is treated with telaglenastat (CB-839) HCl. These potential risks may also apply to TMZ.
* Adolescent patients who require sedation for magnetic resonance imaging (MRI) or magnetic resonance spectroscopy (MRS).
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* The primary language of communication for the patient must be English (dose expansion cohort only). The intended neurocognitive tests have not been validated in patients who do not primarily speak English.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) | Up to 6.5 weeks
  MTD is defined as the dose level below the lowest dose that induces dose limiting toxicity (DLT) in at least 2 patients (out of 6). A total of 6 patients must be treated at the MTD. It is possible that the MTD will be unknown after this study (e.g., if the highest tested dose has fewer than 2 patients with DLT, out of 6). In this case, the highest dose is defined as the RP2D. A 3 + 3 cohort expansion design to determine toxicity-based dose escalation of telaglenastat (CB-839) hydrochloride (HCl) and external beam fractionated radiation therapy (RT) with concurrent temozolomide (TMZ) among patients with IDH-mutated diffuse astrocytoma (DA) or anaplastic astrocytoma (AA).

SECONDARY OUTCOMES:
Objective response rate (ORR) as defined by Response Assessment in Neuro-Oncology (RANO) criteria | Up to 6 months from the start of study treatment
  ORR is defined as the rate of either complete response (CR), partial response (PR), or minor response (MR) by RANO criteria for low-grade gliomas at 6 months after initiation of RT/TMZ/telaglenastat (CB-839) HCl therapy. The ORR will be estimated using properties of the binomial distribution. 95% exact confidence intervals will also be calculated.
Clinical benefit rate (CBR) as defined by RANO criteria | Up to 6 months from the start of study treatment
  CBR is defined as the rate of either CR, PR, MR, or stable disease (SD) by RANO criteria for low-grade gliomas at 6 months after initiation of RT/TMZ/telaglenastat (CB-839) HCl therapy. The CBR will be estimated using properties of the binomial distribution. 95% exact confidence intervals will also be calculated.
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) | Up to 2 years
  The safety and tolerability of RT/TMZ/telaglenastat (CB-839) HCl in patients is based on physician reported adverse event (AE) data.
Progression-free survival (PFS2) as defined by response assessment in neuro-oncology (RANO) criteria | Up to 2 years
  PFS2 rate will be estimated using properties of the binomial distribution. 95% exact confidence intervals will also be calculated.
Overall survival (OS2) as defined by RANO criteria | Up to 2 years
  OS2 rate will be estimated using properties of the binomial distribution. 95% exact confidence intervals will also be calculated.
Assessment of pharmacokinetic (PK) parameters | Pre-dose, 0.5, 1, 2, 4, and 8 hours post-dose on days -7, 1, and 15
  The PK of telaglenastat (CB-839) HCl will also be summarized using descriptive statistics and will be compared to historical data. Measurement of plasma concentrations of telaglenastat (CB-839) HCl and its metabolites (if authentic standards are available) will be performed using validated liquid chromatography-tandem mass spectrometry (LC/MS/MS) assays. The plasma concentration-time data will be analyzed by standard noncompartmental analysis using the program Phoenix WinNonlin 6.4 to determine apparent total clearance of the drug from plasma after oral administration (Cl/F), area under the plasma concentration-time curve from time zero to time t (AUCt), area under the plasma concentration-time curve from time zero to infinity, Cmax, time to reach maximum plasma concentration following drug administration (Tmax), t1/2, and accumulation.
Assessment of self-reported symptoms as measured by MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) instrument | Up to 2 years
  MDASI-BT instrument is used to measure self-reported symptom severity and interference with daily activities. The study will use descriptive statistics to describe how patients rate symptom severity and interference with function at each time point. Compliance rates will be calculated as the number of received valid forms over the number of expected forms. Differences between groups in compliance will be tested by use of Fisher's exact test at every time point.
Assessment of neurocognitive impact | Baseline up to 2 years
  For each test in the battery, a standard error of measurement will be used to derive the Reliable Change Index (RCI) which will be used to represent the 90% confidence interval for the difference in raw scores from baseline to follow-up assessment will be coded as 1 (deterioration), 2 (no change), and 3 (improved) according to the RCI. Percentage of patients in each dose cohort who show meaningful losses or gains in the various tests or test domains over the course of the study will be provided by frequency tables. Dose cohort differences will be compared using chi-squared analysis. Time-to-progressions will be estimated by Kaplan-Meier method and analyzed by Cox regression model adjusting all stratification factors.
Assessment of plasma oncometabolites | Baseline up to day 71
  Plasma oncometabolites (asparagine, aspartate, glutamine, glutamate, and 2-HG) will be compared using changes in values after treatment with the patient's individual baseline values using either the paired t-test or the Mann-Whitney nonparametric U-test as needed. A significant change is defined as a 10% change from baseline.
Assessment of tumor oncometabolites as measured by magnetic resonance spectroscopy (MRS) | Baseline up to day 45
  Tumor oncometabolites (2-HG, glutamine, and glutamate, as measured by MRS) will be compared using changes in values after treatment with the patient's individual baseline values using either the paired t-test or the Mann-Whitney nonparametric U-test as needed. A significant change is defined as a 10% change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sani H Kizilbash, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (25):
- United States (25):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia